CLINICAL TRIAL: NCT04131478
Title: Relationship Between TNF Alpha Gene Polymorphisms and the Pathogenesis of Cachexia in Cancer Patients Treated With Chemotherapy
Brief Title: Effect of Gene Polymorphisms on the Pathogenesis of Cancer Cachexia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Misr International University (Other); Ain Shams University (Other)
Responsible Party: Principal Investigator, Samira Saleh Mostafa, Professor of Pharmacology, Cairo University
Other Study IDs: PT (2387)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Cancer Cachexia
Keywords: cancer cachexia; TNF alfa; pharmacogenetics; mi-RNA
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A heparinized blood sample (5 mls) will be withdrawn from all patients, and divided in 2 aliquots. One aliquot will be spared for DNA and the other for RNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cachectic lung, pancreas, or colon cancer patients.
  Interventions: Genetic: Pharmacogenetic testing
- Control: Non- cachectic lung, pancreas, or colon cancer patients.
  Interventions: Genetic: Pharmacogenetic testing

INTERVENTIONS:
Genetic: Pharmacogenetic testing — Pharmacogenetic testing for TNF alfa

SUMMARY:
Cachexia not only directly increases the morbidity and mortality, it also aggravates the side effects of chemotherapy and reduces the overall quality of life that is often considered the major and direct cause of morbidity of a large proportion (>40%) of cancer patients. Individuals with upper gastrointestinal tumors have the highest rate of developing cachexia associated complications. Chemical and physical signals render an environment conducive for disuse and untenable for proper muscle function leading to wasting.

Till now, several functional single-nucleotide polymorphisms (SNPs) within TNF-α gene have been identified and described as cancer related genetic alterations.

DETAILED DESCRIPTION:
Cachexia is a devastating syndrome that is observed in the majority of end stage cancer patients. Primary symptoms of cancer cachexia comprise of progressive loss in weight and exhaustion of host skeletal muscle tissue as well as adipose tissue reserves.

Cancer cachexia is defined as a multifactorial syndrome, characterized by anorexia as well as diminished body weight, loss of skeletal muscle, and atrophy of adipose tissue (Fearon et al., 2011). Specifically, weight loss of more than 5% over 6 months span in previously healthy individuals or more than 2% in subjects with depletion of current body weight (BMI less than 20 kg/m2) or in individuals with reduced appendicular muscle index (males less than 7.26 kg/m2 and females less than 5.45 kg/m2) constitute the diagnosis of cancer cachexia.

Among potential mechanisms involved in the development of cachexia, the primary initial process is probably the systemic inflammatory response followed by increased production of pro-inflammatory cytokines, such as TNF-α. Multiple biological activities of TNF-α were found in numerous physiological states, including the regulation of cell differentiation, proliferation, apoptosis and metabolism .

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical diagnosis of cancer (eg, lung, pancreas, gastric, biliary, small intestine, or colorectal) Locally, advanced or metastatic cancer scheduled for the first line cytotoxic chemotherapy were eligible for inclusion. Patients who were starting or continuing chemotherapy at the time of screening for participants
* The duration was set based on standard period of first line chemotherapy
* Age of 18 years to 80 years
* Written informed consent of the subject to participate in the study

Exclusion Criteria:

* Planned to have surgical procedures at the time of recruitment
* Underwent surgery during the study or in the month prior to the study and did not have chemotherapy scheduled postsurgery
* Had any comorbidities that could affect the interpretation of study findings (eg, HIV, AIDS, Alzheimer's disease, movement disorder, acute myocardial infarction within last 3 months, hepatitis)
* Had open burn sites or infected wounds
* Were diagnosed with esophageal cancer with a swallowing difficulty in mechanical nature
* Had an uncorrected, mechanical digestive obstruction
* Pregnant or nursing women
* Disorders associated with change in micro RNA (miR-155) level (Rheumatic Arthritis, Osteoarthritis, Atopic Eczema, Down Syndrome, Breast cancer, Endometrioid adenocarcinoma, AML, CLL, PC thyroid tumors)
* Inflammatory and autoimmune diseases (Multiple Sclerosis, Psoriasis and Systemic Lupus Erythematous)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cachectic and non- cachectic cancer patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-20 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
TNF-α -1031T/C and 308 G/A | 6 months
  To detect the incidence of tumor necrosis factor (TNF-α -1031T/C and 308 G/A) gene polymorphism in the Egyptian cancer patients with local/advanced or metastatic cancer and investigation of TNF-α -1031T/C and 308 G/A as a cachexia risk factor.

SECONDARY OUTCOMES:
Biochemical markers | 6 months
  SOCS1, TAB2 and FOXP3

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No